CLINICAL TRIAL: NCT01992796
Title: Phase III Study of Irbersartan for the Early Treatment of Severe Sepsis Patients
Brief Title: Angiotensin II Antagonist in Severe Sepsis
Acronym: SartSep
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Salerno (Other)
Collaborators: Federico II University (Other)
Responsible Party: Principal Investigator, Ornella Piazza, Reasercher, University of Salerno
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FARM97AJNN
Record Dates: First submitted 2013-11-11; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Severe Sepsis
Keywords: irbesartan, angiotensin, sepsis
MeSH Terms: conditions — Sepsis | interventions — Irbesartan; candesartan; Telmisartan; olmesartan; Valsartan

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- irbesartan (Experimental): Irbesartan (total dose of 75 mg) or placebo administered every 24 hrs for 15 days. Moreover, the sepsis management will follow standard international guidelines (Crit Care Med.2008 Jan;36(1):296-327. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock).
  Duration of treatment: Irbesartan 75 mg daily for 15 days; only one cycle. Follow up will last 90 days both for treatment and control arm.
  * Route of administration : oral by nasogastric tube.
  * Medication permitted and not permitted during the trial:
  all the therapeutic interventions for sepsis management as indicated by international guidelines are admitted. During the trial are not permitted: ACE inhibitors, ARBs different from Irbersartan, angiotensin I synthesis inhibitors
  Interventions: Drug: Irbesartan
- Placebo (Placebo Comparator): Packaging and labelling for blinding purposes: tablets of placebo looking like the study drug

INTERVENTIONS:
Drug: Irbesartan — 75 mg/per os/for 15 days
  Other Names: Candesartan.; Telmisartan.; Olmesartan.; Lortaan; Losaprex; Neolotan; Tevetenz; Rixil; Tareg; Valpression; Aprovel; Karvea.
  Arms: irbesartan

SUMMARY:
The investigators propose a clinical study of irbersartan for the early treatment of severe sepsis patients with elevated predicted risk of death between. This study will evaluate whether early administration of the the angiotensin receptor blocker irbersartan provides significant reduction of 28 days mortality and multi organ failure incidence to patients with severe sepsis.

DETAILED DESCRIPTION:
Background: Angiotensin II (ANG II) is a potent vasoconstrictor and diminishes vasodilator responses in arteries. In addition to direct effects on vascular tone, ANG II affects multiple aspects of microvascular function through promotion of leukostasis, induction of capillary permeability and depletion of glutathione. Binding of ANG II to its receptors (in particular AT1) mediates intracellular free radical generation that contributes to tissue damage by promoting mitochondrial dysfunction.

Angiotensin receptor blockers (ARBs) interrupt renin-angiotensin system (RAS) overactivity by blocking a specific receptor that mediates the pathogenic activity of angiotensin II. Objectives: The clinical question objective of this study is if the antiinflammatory effect of ARBs is relevant in sepsis management and in particular if ARBs are able to improve survival and reduce the incidence of Multi Organ Failure in septic patients.

Methods:

STUDY DESIGN: Experimental; prospective, randomized, multicenter, phase III trial.

STUDY POPULATION: Three hundred adults within 12 hrs of recognition of severe sepsis, with Acute Physiology and Chronic Health Evaluation (APACHE) II-predicted risk of mortality between 20% and 80% are eligible.

Settings: 5 Italian Intensive Care Units. Oral irbesartan (total dose of 75 mg) or placebo administered every 24 hrs for 15 days. Analysis of data performed by a blind operator. Expected results: about 25% reduction in 28-day mortality rate and incidence of multi organ failure in the study population.

ELIGIBILITY:
Inclusion Criteria: adults within 12 hrs of recognition of severe sepsis, with Acute Physiology and Chronic Health Evaluation (APACHE) II-predicted risk of mortality between 20% and 80% are eligible.

Exclusion Criteria:Patients already treated with ACE inhibitors or ARBs will be excluded. Patients admitted in shock conditions (systolic blood pressure lower than 90 mmHg) will be excluded. Patients with severe renal failure (serum creatinine of 2.0 mg/dL or dialysis) will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
mortality | 28 days

SECONDARY OUTCOMES:
Incidence of altered organ function in sepsis patients measured by SOFA score (Sequential Organ Failure Assessment score) | 28 day
  Incidence of altered organ function in sepsis patients measured by SOFA score (Sequential Organ Failure Assessment score). It is known that respiratory failure is more common in the first 72 hours after the original insult, hepatic failure after 5-7 days, gastrointestinal bleeding within 10-15 days and renal failure in 11-17 days: the SOFA score will be checked every day for 28 days. The SOFA score is a scoring system to determine the extent of a person's organ function or rate of failure. The score is based on six different scores, one each for the respiratory, cardiovascular, hepatic, coagulation, renal and neurological systems.
  Creatinine serum levels, bilirubin, coagulation tests, blood gases and neurological clinical evaluation will be performed every day for the first 15 days; they will be retested at least once a week and at the end of the study protocol (28-day).

OTHER OUTCOMES:
Incidence of renal failure | 28 days
  Creatinine (mg/dl) (SOFA score) 1.2 - 1.9 (1) 2.0 - 3.4 (2) 3.5 - 4.9 (or urine output< 500 ml/d) (3) > 5.0 (or urine output< 200 ml/d) (4)

CONTACTS AND LOCATIONS:
Overall Officials: Rosalba Tufano, MD, Study Director — Federico II University
Locations (1):
- Università di Salerno, Salerno, Italy